CLINICAL TRIAL: NCT02646436
Title: Peritoneal Dialysis as an Option of Unplanned Initiation of Chronic Dialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Dayana Bitencourt Dias, Medical nephrologist, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UEPJMF
Record Dates: First submitted 2015-12-15; First posted 2016-01-05 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Disorders Associated With Peritoneal Dialysis
Keywords: unplanned peritoneal dialysis; unplanned heamodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HD treatment (Other): Patients with absolute contraindication to the PD method - presence of recent abdominal surgery (less than 30 days); multiple previous abdominal surgery (more than two); presence of fibrosis or peritoneal adhesions; fungal peritonitis; severe respiratory insufficiency (FiO2> 70%); abdominal infections; severe hyperkalemia with changes characteristic in EKG; and acute pulmonary edema - will be treated with HD.
  Interventions: Other: HD treatment
- PD treatment (Other): Patients stage 5 (creatinine clearance < 15 ml/min) requiring dialysis treatment immediately without absolute contraindication to the PD method will receive unplanned PD treatment. High volume PD (HVPD) will be used during the first 7 days of PD in order to achieve metabolic and fluid control. The procedure for acute PD has been published recently by our team . At this point, patients will be discharged from hospital and they will be treated by intermitent PD at the dialysis unit of the University Hospital.until their family be trained and home be prepared for the implementation of technique.
  Interventions: Other: PD treatment

INTERVENTIONS:
Other: HD treatment — Patients with absolute contraindication to the PD method will be treated with HD. HD will be performed after implantation of central venous catheter using Seldinger technique by nephrology team.
  Arms: HD treatment
Other: PD treatment — Patients without absolute contraindication to the PD method will be treated with PD. PD will be performed after implantation of peritoneal catheter using Seldinger technique by nephrology team.
  Arms: PD treatment

SUMMARY:
Peritoneal dialysis (PD) has become a well-established complementary alternative to haemodialysis (HD) as first-line renal replacement modality. At department of Botucatu Medical School, more than 60% of the chronic kidney disease (CKD) stage 5 patients are started urgently on chronic dialysis due to late referral or unexpected deterioration of residual renal function. These patients, although suitable for PD, were previously started on HD using central venous catheter. Since July 2014 patients have been offered urgent start on chronic PD right after PD-catheter insertion by percutaneous surgery, using Seldinger technique. The main objective is to compare technique and patients survival on unplanned PD vs. unplanned HD in the first 180 days. Methodology: Quasi experimental study which will describe how acute PD will initiated using high volume PD until metabolic and fluid control right after (<48 h) PD catheter placement standard prescription for a 12 h overnight automatic PD until hospital discharge and intermittent PD at dialysis unit family training.

DETAILED DESCRIPTION:
1. Background:

   Chronic Kidney Disease (CKD) is a matter of global public health. Data from United States of America (USA) has shown a steady increase in the number of patients on renal replacement therapy (RRT). The census of the Brazilian Society of Nephrology (SBN) showed 65,121 patients on dialysis program in 2005, while in 2011 there were 91,314 and in 2013, there were more than 100,000 patients on dialysis in Brazil.

   Among the methods of dialysis, nephrologists have two options: the peritoneal dialysis (PD) and hemodialysis (HD), which is the most commonly used method in the world. Although, historically, PD was widely used in nephrology, for not clear reasons it has been underutilized in last years, especially in incident patients on RRT. In Brazil, data from 2013 showed that 90.6% of chronic patients underwent HD and only 9.4% were treated by PD.

   Several studies have compared the differences between the two types of dialysis - PD vs. HD - in incident patients on RRT. There is no evidence of the superiority of one method over the other in regards to general mortality within the first two years of therapy.

   Recently, some authors have pointed out the impact of the vascular access used in the mortality of incident patients in HD. These studies found that central venous catheters (CVC) use is associated with reduced survival, especially in the first 90 days of RRT. Furthermore, there is a greater risk of bacteremia, sepsis and hospitalizations in patients using CVC when compared to patients using arteriovenous fistulas (AVF) or graft or PD.

   In this scenario, the PD appears as an option of unplanned initiation of chronic dialysis. Starting dialysis in an unplanned manner is a frequent situation in dialysis centre even for patients without or with a regular nephrology follow-up.

   Unplanned dialysis initiation can be defined as an end-stage renal disease patient beginning HD with no functional vascular access, using CVC or as the starting PD in less than 7 days after peritoneal catheter implantation. It has been shown that unplanned dialysis and using temporary HD catheters are independently associated with mortality in incident dialysis patients. For no clear reasons, PD is underused in unplanned dialysis patients.

   In Brazil, approximately 60% of incident patients on RRT have no definitive access and need to be treated through CVC.

   However, there are few studies that describe PD method as an immediate treatment option in patients without functioning vascular access and only two small studies that compared unplanned start of HD vs. PD.

   Lobbedez et al followed by the 2-year period, 60 patients who started unplanned dialysis - 34 patients treated by PD and 26 by HD. Among the patients who started on PD, no significant difference in mechanical or infectious complications when compared to patients who had "rest time" post-catheter insertion. There was no significant difference between the two unplanned dialysis methods (HD x DP) in patients survival (78.8% in the HD group vs. 82.9% in PD (p = 0.26). After adjusting for comorbidities index, survival between the two groups remained similar.

   Koch et al. evaluated 57 incident patients in unplanned HD and 66 in unplanned PD. HD patients had more bacteremia than PD patients in the first 6 months of dialysis (21.1% vs 3%, p <0.01), which was associated with the use of CVC as initial access . However, there was no significant difference in the mortality rates between the two methods.

   So it is clearly needed to show that PD is a suitable method for unplanned dialysis patients and that acute automated PD may help nephrologists to deal with patients without any permanent vascular access at dialysis initiation. The investigators believe that PD can offer the advantage of not using CVC, which can reduce the morbidity and mortality of CKD patients. In addition, in October/2014, there was not vacancy for incident patients on chronic HD in Dialysis Unit of University Hospital of Botucatu Medical School, worrying fact for a high complexity service that has received an average of 8 incident patients on RRT, monthly.
2. Objectives:

   The main objective of this study is to compare technique and patients survival on unplanned PD vs. unplanned HD in the first 180 days of therapy.

   This study is also carried out:
   * To compare the rates of hospitalization and infectious related with PD vs HD.
   * To determine the impact on the PD and HD programs (growing or reduction)
3. Methodology 3.1. Patients: This study is a quasi experimental study that will evaluate incident unplanned PD and HD patients at Dialysis Unit of Botucatu Medical School. In an attempt to increase the use of PD for unplanned dialysis patients, a programme devoted to this group of patients has been set up since 1 November 2014.

Inclusion criteria are CKD patients stage 5 (creatinine clearance < 15 ml/min) requiring dialysis treatment immediately. Unplanned HD was defined as initiation without definitive vascular access and using CVC and unplanned PD as initiation in less than 48 hours after implantation of the peritoneal catheter.

Absolute contraindication to the PD method are: presence of recent abdominal surgery (less than 30 days); multiple previous abdominal surgery (more than two); severe respiratory insufficiency (FiO2> 70%); abdominal infections; severe hyperkalemia with changes characteristic in EKG; and acute pulmonary edema. These patients will be treated with HD.

The decision concerning the dialysis modality has been made according to the medical's indications and patient's choice. The implant of Tenckhoff catheter will be held through the percutaneous Seldinger technique by nephrology team. High volume PD (HVPD) will be used during the first 7 days of PD in order to achieve metabolic and fluid control. The procedure for acute PD has been published recently. When HD is the modality of choice, a temporary catheter is inserted rapidly by nephrologist, at the bedside if necessary, and after one week it will be changed to tunneled line.

Patients will be followed by the same research team from the time of the peritoneal catheter implantation until the outcome (stay in the method for a minimum period of 90 days, death, transplantation, recovery of renal function or switch to HD due to technical failure or infectious and mechanical complications without success with the treatment).

3.2. Research Protocol: The study protocol will consist of clinical and laboratory data, dialysis and monitoring of patients on PD and HD unplanned.

3.2.1. General data:

* Identification: name, gender, age, color
* Etiology and stage of CKD
* Presence of co-morbidities
* Start of unplanned dialysis (date)
* Date of the peritoneal catheter or CVC implantation
* Complications during or after implantation of the catheter
* Start date of family training (PD method)
* Date of the end of the family training (PD method)
* Number of training days (PD method)

3.2.2. Dialysis:

• Dialysis indications

PD: Catheter implantation using the Seldinger technique

* Prescription: HVPD to achieve adequate metabolic and fluid control. At this point, patient will be discharged from hospital.
* Intermitent PD on alternate days or daily: patients will be treated by PD at the dialysis unit of the University Hospital every other day or every day, according to their lab exams and clinic exam. Laboratorial exams will be performed weekly, until their family be trained and home be prepared for the implementation of technique.

HD: on alternate days at Dialysis Unit

3.2.3. Follow up of unplanned dialysis patients:

* Evaluation of mechanical and infectious complications related to PD or HD
* Technique and patients survival

3.3. Statistical Analysis: The sample size calculation was based on the assumption the difference of 15% between patients undergoing unplanned PD and HD in outcomes as hospitalization, infection and mortality. With a first-order error of 5% and a power of 80% a sample size of 94 patients is needed in each treatment group.

From the study protocol, the data will be entered in a spreadsheet and verified typographical errors and their analysis will be performed using the statistical program SAS for Windows (version 9.2: SAS Institute,Cary, NC, USA, 2012). Initially descriptive analysis will be done for all patients treated in the period, calculated measures of central tendency and dispersion for continuous variables and frequencies for categorical variables. Patients will be separated into two groups according to initiation modality (unplanned PD group and unplanned HD group) in order to evaluate the impact of unplanned PD on technique and patient survival and on survival free of peritonitis. Intent-to-treat analysis will be used to analyse patient survival. T-test will be used to compare parametric continue variables between the two groups and Kruskal-Wallis test for nonparametric continue variables. Chi Square will be used to compare categorical variable between the two groups. For the analysis of repeated measures, asymmetric distribution (gamma) under the GENMOD procedure will be used.

At the end of the study will be presented survival curves using Kaplan Meyer of patients and the method during the monitoring period. Cox proportional hazards model was used to adjust survival on baseline characteristics. The statistical difference was considered to be significant for p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are CKD patients stage 5 (creatinine clearance < 15 ml/min) requiring dialysis treatment immediately.

Exclusion Criteria:

* Presence of recent abdominal surgery (less than 30 days)
* Multiple previous abdominal surgery (more than two)
* Severe respiratory insufficiency (FiO2> 70%)
* Abdominal infections
* Severe hyperkalemia with changes characteristic in EKG
* Acute pulmonary edema.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2014-11-30; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Comparasion of patients survival between unplanned PD vs. unplanned HD | 180 days
  The main objective of this study is to compare patients survival on unplanned PD vs. unplanned HD in the first 180 days of therapy

SECONDARY OUTCOMES:
Comparasion of hospitalization between unplanned PD vs. unplanned HD | 180 days
  To compare rates of hospitalization (%) between unplanned HD vs. unplanned PD
Comparasion of mechanical complications (%) between unplanned PD vs. unplanned HD | 180 days
  To compare mechanical complications (%) between unplanned HD vs. unplanned PD
Comparasion of infectious complications (%) between unplanned PD vs. unplanned HD | 180 days
  To compare infectious complicatios (%) between unplanned HD vs. unplanned PD

OTHER OUTCOMES:
Evaluate the increase of PD penetration rate among incident patients initiating chronic dialysis therapy (%) | Two years
  To evaluate the impact on growing of PD chronic program (%)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela ponce, Study Director — Botucatu Medical School
Locations (1):
- Paulista State University "Júlio de Mesquita Filho", Botucatu, São Paulo, Brazil

REFERENCES:
- [Background] Ponce D, Buffarah MB, Goes C, Balbi A. Peritoneal Dialysis in Acute Kidney Injury: Trends in the Outcome across Time Periods. PLoS One. 2015 May 12;10(5):e0126436. doi: 10.1371/journal.pone.0126436. eCollection 2015. PMID 25965868
- [Background] Pajek J. Overcoming the Underutilisation of Peritoneal Dialysis. Biomed Res Int. 2015;2015:431092. doi: 10.1155/2015/431092. Epub 2015 Nov 11. PMID 26640787
- [Background] Ivarsen P, Povlsen JV. Can peritoneal dialysis be applied for unplanned initiation of chronic dialysis? Nephrol Dial Transplant. 2014 Dec;29(12):2201-6. doi: 10.1093/ndt/gft487. Epub 2013 Dec 17. PMID 24353321
- [Background] Lecouf A, Ryckelynck JP, Ficheux M, Henri P, Lobbedez T. A new paradigm: home therapy for patients who start dialysis in an unplanned way. J Ren Care. 2013 Jan;39 Suppl 1:50-5. doi: 10.1111/j.1755-6686.2013.00336.x. PMID 23464914
- [Background] Koch M, Kohnle M, Trapp R, Haastert B, Rump LC, Aker S. Comparable outcome of acute unplanned peritoneal dialysis and haemodialysis. Nephrol Dial Transplant. 2012 Jan;27(1):375-80. doi: 10.1093/ndt/gfr262. Epub 2011 May 28. PMID 21622993
- [Background] Korevaar JC, Feith GW, Dekker FW, van Manen JG, Boeschoten EW, Bossuyt PM, Krediet RT; NECOSAD Study Group. Effect of starting with hemodialysis compared with peritoneal dialysis in patients new on dialysis treatment: a randomized controlled trial. Kidney Int. 2003 Dec;64(6):2222-8. doi: 10.1046/j.1523-1755.2003.00321.x. PMID 14633146
- [Background] Vonesh EF, Snyder JJ, Foley RN, Collins AJ. Mortality studies comparing peritoneal dialysis and hemodialysis: what do they tell us? Kidney Int Suppl. 2006 Nov;(103):S3-11. doi: 10.1038/sj.ki.5001910. PMID 17080109
- [Background] Chaudhary K, Sangha H, Khanna R. Peritoneal dialysis first: rationale. Clin J Am Soc Nephrol. 2011 Feb;6(2):447-56. doi: 10.2215/CJN.07920910. Epub 2010 Nov 29. PMID 21115629
- [Background] Perl J, Wald R, McFarlane P, Bargman JM, Vonesh E, Na Y, Jassal SV, Moist L. Hemodialysis vascular access modifies the association between dialysis modality and survival. J Am Soc Nephrol. 2011 Jun;22(6):1113-21. doi: 10.1681/ASN.2010111155. Epub 2011 Apr 21. PMID 21511830
- [Background] Heaf JG, Lokkegaard H, Madsen M. Initial survival advantage of peritoneal dialysis relative to haemodialysis. Nephrol Dial Transplant. 2002 Jan;17(1):112-7. doi: 10.1093/ndt/17.1.112. PMID 11773473
- [Result] Liu FX, Ghaffari A, Dhatt H, Kumar V, Balsera C, Wallace E, Khairullah Q, Lesher B, Gao X, Henderson H, LaFleur P, Delgado EM, Alvarez MM, Hartley J, McClernon M, Walton S, Guest S. Economic evaluation of urgent-start peritoneal dialysis versus urgent-start hemodialysis in the United States. Medicine (Baltimore). 2014 Dec;93(28):e293. doi: 10.1097/MD.0000000000000293. PMID 25526471
- [Derived] Htay H, Johnson DW, Craig JC, Teixeira-Pinto A, Hawley CM, Cho Y. Urgent-start peritoneal dialysis versus conventional-start peritoneal dialysis for people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 15;12(12):CD012913. doi: 10.1002/14651858.CD012913.pub2. PMID 33320346